CLINICAL TRIAL: NCT06407271
Title: Effect of Abutment 3-dimensional Configuration on Peri-implant Soft and Hard Tissue in the Esthetic Zone - Randomized Clinical Trial
Brief Title: Effect of Abutment Configuration on Peri-implant Soft and Hard Tissue in the Esthetic Zone - Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 260/2023
Record Dates: First submitted 2024-04-12; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-12

CONDITIONS: Dental Implants, Single-Tooth; Dental Implant-Abutment Design
Keywords: Peri-Implant Tissue Management; CAD-CAM; Dental Implants, Single-Tooth; Dental Implant-Abutment Design

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD/CAM custom ZrO2 healing abutment (Experimental): Application of custom, zirconium-dioxide healing abutment, fabricated with computer aided design and manufacturing, following immediate implantation.
  Interventions: Device: CAD/CAM custom ZrO2 healing abutment
- Cylindrical ZrO2 healing abutment (Active Comparator): Application of cylindrical, zirconium-dioxide healing abutment following immediate implantation.
  Interventions: Device: Cylindrical ZrO2 healing abutment

INTERVENTIONS:
Device: CAD/CAM custom ZrO2 healing abutment — Application of custom, zirconium-dioxide healing abutment, fabricated with computer aided design and manufacturing, following immediate implantation.
  Other Names: CAD-CAM custom zirconium-dioxide healing abutment
  Arms: CAD/CAM custom ZrO2 healing abutment
Device: Cylindrical ZrO2 healing abutment — Application of cylindrical, zirconium-dioxide healing abutment following immediate implantation.
  Other Names: Cylindrical zirconium-dioxide healing abutment
  Arms: Cylindrical ZrO2 healing abutment

SUMMARY:
The aims of our study are to investigate in patients with immediate implantation replacing a single tooth in the maxillary anterior (#FDI 15-25) region the effect of (a) custom vs cylindrical stock healing abutments, then (b) screw retained single ceramic crowns, on the peri implant hard- and soft-tissue formation and blood flow.

DETAILED DESCRIPTION:
AIMS:

In the maxilla, in the aesthetic zone, in patients with a thick phenotype, for a crown anchored with a solo immediate implant:

I.A To investigate hard and soft tissue volume changes around custom CAD/CAM (computer-aided design and manufacturing) vs. cylindrical zirconiom-dioxide (ZrO2) healing abutments 4 months after their fixation for immediate implant placement.

I.B To measure the thickness of keratinized mucosa by ultrasound I.C Monitoring microcirculation in wound healing by laser speckle contrast imaging (LSCI) and ultrasound.

II. Custom zirconia abutment (on Ti-base) retained, screw-retained all-ceramic solo restorations:

* Evaluation of hard and soft tissue volume changes
* Esthetic evaluation (Pink and White Aesthetic Scores (PES, WES)), FIPS (functional implant prosthodontic score), pain, follow-up of biological and technical complications at 1 and 3 years.

ARMS:

A. immediate implantation + cylindrical healing abutment + CAD/CAM screw-retained (on Ti-base), full-countour monolithic zirconium-dioxide restoration

B. immediate implantation + custom healing abutment + CAD/CAM screw-retained (on Ti-base), custom ZrO2 abutment retained all-ceramic restoration with hand-built-up supramucosal veneering

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years
* good general health
* good oral hygiene (FMPS < 25%)
* healthy periodontium (PPD < 4mm)
* thick phenotype
* maxilla anterior region (extended to 15-25 positions)
* solo missing teeth, intact adjacent teeth
* type 1 alveolar shape after extraction 1
* retained occlusion
* baseline buccal bone wall thickness at least 1.5 mm, based on intact CBCT scan
* patient voluntarily accepts and signs the information and consent form for the study

Exclusion Criteria:

* general ill health
* general surgical or oral surgery contraindication
* a patient who has undergone local radiotherapy
* active periodontal inflammation, inflammation of the alveolar cavity
* smoking
* posterior region
* pregnancy, lactation
* psychological or mental involvement affecting individual plaque control
* presence of an implant adjacent to the planned implant
* inadequate oral hygiene
* need for vertical bone augmentation
* gingival recession
* Inappropriate implant position for screw fixation
* bruxism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
midfacial keratinized mucosa volume | 4, 12, 36 months post op.
  Volume changes in midfacial mucosa [mm]
midfacial keratinized mucosa width | 4, 12, 36 months post op.
  Keratinized mucosa width [mm]
Keratinized mucosa thickness | before implantation, 4,12, 36 months post op.
  Keratinized mucosa thickness with ultrasound [mm]

SECONDARY OUTCOMES:
soft tissue volume | 4, 12, 36 months post op.
  Follow-up of 2D linear and 3D volumetric changes in soft tissue using intraoral scanner
laser speckle contrast imaging (LSCI) | at 0-7., 0., 1., 4., 7., 14. day, and 1., 2., 4., 6., 12 month after implantation
  blood flow measurement with laser speckle contrast imaging
ultrasound | at 0-7., 0., 1., 4., 7., 14. day, and 1., 2., 4., 6., 12 month after implantation
  blood flow measurement with ultrasound
marginal bone loss | 4, 12, 36 months post op.
  marginal bone loss
Implant survival | 4, 12, 36 months
  Number of survived implants out of total implants placed
full mouth plaque score (FMPS) | 0., 1., 7., 14. day, and 1., 2., 4., 6., 12., 36. month after implantation
  % of sites with dental plaque over total measures sites
full mouth bleeding score (FMBS) | 0. day, and 4., 12., 36. month after implantation
  % of sites with bleeding over total measures sites
Probing depth (PPD) | 0., 4., 12., 36. month after implantation
  Probing pocket depth
Functional implant prosthodontic score (FIPS) | 4 months after implantation, at final restoration delivery
  Functional implant prosthodontic score
Pain at delivery | 4 months after implantation, at final restoration delivery
  Pain numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Krisztina Mikulás, PhD, Principal Investigator — Semmelweis University, Department of Prosthodontics
Locations (1):
- Semmelweis University, Department of Prosthodontics, Budapest, Pest County, Hungary